CLINICAL TRIAL: NCT01457001
Title: Controlled Randomised Interventional Trial on the Use of 25-OH D Vitamin in Haemodialysis Patients.
Brief Title: Clinical Trial on the Use of 25-OH -D Vitamin in Haemodialysis Patients
Acronym: NUTRIVITA-D001
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Italian Society of Nephrology (Other)
Collaborators: Società Italiana di Nefrologia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NUTRI-VITA-D001
Record Dates: First submitted 2011-10-13; First posted 2011-10-21 (Estimated); Last update posted 2016-12-01 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Renal Failure
Keywords: chronic haemodialysis; 25-OH-D vitamin
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 25-OH-D vitamin (Experimental)
  Interventions: Drug: 25-OH-D vitamin
- control (No Intervention)

INTERVENTIONS:
Drug: 25-OH-D vitamin
  Arms: 25-OH-D vitamin

SUMMARY:
Multicentric randomized Italian clinical trial, open label, not for profit. To evaluate the efficacy of 25-OH-D vitamin in terms of myocardial infarction, stroke, sudden death, death for other causes in chronic haemodialysis patients. Two arms of treatment: 25-OH-D vitamin per os versus no treatment.

ELIGIBILITY:
Inclusion Criteria:

* age >= 18 years
* hematic PTH level twofold-ninefold the upper limit
* hematic level of 25-OH-D vitamin < 30 ng/ml

Exclusion Criteria:

* renal transplant or peritoneal dialysis less than 3 years ago
* pregnancy
* breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2012-11; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Vital status | During the follow up, every three months for three years
  Death for all causes but traumatic.
Onset of non fatal myocardial infarction | During the follow up, every three months for three years
  Cumulative with the vital status
Onset of non fatal stroke | During the follow up, every three months for three years
  Cumulative with the vital status

SECONDARY OUTCOMES:
fatal myocardial infarction | During the follow up, every three months for three years
non fatal myocardial infarction | During the follow up, every three months for three years
fatal stroke | During the follow up, every three months for three years
non fatal stroke | During the follow up, every three months for three years
sudden death | During the follow up, every three months for three years
death for other causes (not traumatic) | During the follow up, every three months for three years
frequency of hypercalcemia (>10.5 mg/dl) | During the follow up, every three months for three years
frequency of hyperphosphoremia (>5.5 mg/dl) | During the follow up, every three months for three years
frequency of normal level of 25-OH-D vitamin (>30 ng/ml) | During the follow up, every three months for three years
frequency of 25-OH-D vitamin >100 ng/ml | During the follow up, every three months for three years
frequency of reduction of therapy with calcitriol and/or paricalcitol and/or calcium mimetics and/or phosphorus chelators | During the follow up, every three months for three years
frequency of parathyroid surgery | During the follow up, every three months for three years

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Morrone, MD, Study Chair — Società Italiana di Nefrologia
Locations (28):
- Italy (28):
  - Ospedale "A. Landolfi", Solofra, Avellino
  - UOC Nefrologia e Dialisi - AO Moscati, Avellino, AV
  - Ospedale Miulli, Acquaviva delle Fonti, Bari
  - Ospedale Umberto I, Altamura, Bari
  - Ospedale Santa Maria degli Angeli, Putignano, Bari
  - U.O.C. Nefrologia e Dialisi - PO Beato Angelico, Acri, CS
  - Presidio Ospedaliero Anagni, Anagni, Frosinone
  - P.O.N.S Bonaria, San Gavino Monreale, Medio Campidano
  - Ospedale Civile di Alghero ASL n°1, Alghero, Sassari
  - Ospedale Civile, Manduria, Taranto
  - P.O. Atri - Asl Teramo, Atri, Teramo
  - SC Nefrologia e Dialisi - Ospedale Martini, Torino, TO
  - Azienda Ospedaliera Gaetano Rummo, Benevento
  - AORN Sant'Anna e San Sebastiano Caserta, Caserta
  - A.O. Istituti Ospedalieri di Cremona, Cremona
  - Ospedale S.Giovanni di Dio, Florence
  - Azienda Ospedaliera Universitaria OO.RR Foggia, Foggia
  - Ospedale ICOT, Latina
  - Università di Messina, Messina
  - Azienda Ospedaliera Ospedali Riuniti Papardo Piemonte, Messina
  - 1° Divisione di Nefrologia - Azienda Universitaria Policlinico, Napoli
  - Reparto di Nefrologia - Ospedale Cardarelli, Napoli
  - Ospedale Santa Maria del Popolo degli Incurabili, Napoli
  - ARNAS "Civico, Di Cristina", Palermo
  - A.O. Ospedali Riuniti Marche Nord-Presidio San Salvatore, Pesaro
  - AO Universitaria Pisana Presidio di Cisanello, Pisa
  - Ospedale G.B Grassi, Roma
  - Ospedale di Belcolle, Viterbo

REFERENCES:
- [Derived] Morrone L, Palmer SC, Saglimbene VM, Perna A, Cianciolo G, Russo D, Gesualdo L, Natale P, Santoro A, Mazzaferro S, Cozzolino M, Cupisti A, Di Luca M, Di Iorio B, Strippoli GFM; Mineral Metabolism Study Group of the Italian Society of Nephrology. Calcifediol supplementation in adults on hemodialysis: a randomized controlled trial. J Nephrol. 2022 Mar;35(2):517-525. doi: 10.1007/s40620-021-01104-z. Epub 2021 Jun 26. PMID 34173940